CLINICAL TRIAL: NCT03033446
Title: A Phase II Open-Label, Single Centre, Non-Randomised Trial Of Y90-Radioembolization In Combination With Nivolumab In Asian Patients With Advanced Hepatocellular Carcinoma
Brief Title: Study of Y90-Radioembolization With Nivolumab in Asians With Hepatocellular Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-678
Record Dates: First submitted 2017-01-18; First posted 2017-01-26 (Estimated); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: HepatoCellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Y90-Radioembolization and Nivolumab (Experimental)
  Interventions: Radiation: Y-90 Radioembolization; Drug: Nivolumab

INTERVENTIONS:
Radiation: Y-90 Radioembolization — Dose of Yttrium-90 is determined based on BSA, size of liver tumor, and dose modifications required for percent lung shunting between 10-20% on the Tc-99MMA scan
  Other Names: Selective Internal Radiation Therapy
Drug: Nivolumab — 21 days after Radioembolization, 240mg of IV Nivolumab over 30 minutes will be administered every 2 weeks
  Other Names: Opdivo

SUMMARY:
The purpose of this study is to evaluate the effect of liver-localised radioembolization and nivolumab on liver cancer.

DETAILED DESCRIPTION:
The hypothesis is that liver-localized radioembolization will stimulate tumour and/or HBV specific T cell responses that are associated with favourable patient outcomes and that can be boosted using nivolumab anti-PD1 checkpoint blockade immunotherapy.

Primary objective

To evaluate the response rates of Y90 radioembolization in combination with nivolumab in HCC

Secondary objectives

1. To evaluate time to response, response duration, time to treatment progression and sites of progression when RE is combined with nivolumab
2. To assess progression free survival and overall survival when RE is combined with nivolumab
3. To assess the quality of life using the FACT-HEP score and EORTC QLQ-C30
4. To assess the safety and tolerability of the combination of RE and nivolumab

Exploratory objectives

1. To evaluate the relationship between tumor biopsy PD-L1 expression and response to treatment with Y90 radioembolization in combination with nivolumab
2. To assess relationship between blood lymphocyte (e.g., T cell) activation and phenotypic profiles with response to treatment with Y90 radioembolization in combination with nivolumab, using mass cytometry and fluorescence flow cytometry.
3. To assess relationship between HCC tumour mutational burden and response to treatment with Y90 radioembolization in combination with nivolumab using whole-exome sequencing of tumour biopsy samples
4. Where possible, to evaluate antigen-specific T cell responses to known HBV, HCC tumour (including candidate mutation-derived tumour neo-antigens) and other unrelated antigens (e.g. CMV, EBV, Influenza) in the blood and to assess kinetic changes in these responses associated with response to treatment with Y90 radioembolization in combination with nivolumab using mass cytometry and fluorescence flow cytometry.

Administration of study drug The first dose of nivolumab will be administered 21 days (+/- 3 days) after completion of RE. [The dose of Yttrium-90 will be determined as per institution norm by the Nuclear Medicine physician, based on factors such as the subject's Body Surface Area (BSA), the size of the tumour within the liver, and any dose modifications required for percent lung shunting between 10 - 20% on the Tc-99MMA scan].

The dose given will be intravenous 240mg absolute over 30 minutes. Subsequent doses of nivolumab will be administered in the outpatient setting at NCCS. After the first dose, intravenous nivolumab 240mg will be given every 2 weeks.

A US or CT guided liver biopsy will be conducted by an interventional radiologist on C1D8 Subjects will be assessed for the following at EVERY visit: physical examination, ECOG status, vital signs, Child-Pugh score and ALBI score CT or MRI scans to assess response to treatment will be done before cycle 4, 8, 12 and then after every 12 weeks thereafter (±7 days).

FACT-HEP and EORTC QLQ C30 version 3.0 questionnaire at cycle 4 and 8.

Follow-Up Visit will be done 2-3 months after last dose. Survival updates will be obtained by phone every 3-4 months after the follow-up visit and any new anti-cancer treatment given to the subject will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with hepatocellular carcinoma (HCC) that is not suitable for resection or liver transplant, who are planned for Y90 radioembolization as per institutional practice.
2. Patients must have measurable disease with target lesion in liver, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan.
3. Diagnosis of HCC confirmed by histology/cytology or clinically by AASLD criteria in cirrhotic subjects. Patients without cirrhosis require histological confirmation of diagnosis
4. No prior Y90 radioembolization therapy. Prior local therapies, such as surgery, hepatic artery embolization/chemoembolization, radiofrequency ablation, percutaneous ethanol injection or cryoabalastion is allowed, if the index lesion(s) remains outside of the treatment field or has progressed since prior treatment. Local therapy must have been completed at least 4 weeks prior to the baseline scan
5. Age ≥ 21 years.
6. ECOG performance status ≤ 2
7. Life expectancy of greater than 3 months
8. Only patients with Child-Pugh score for liver cirrhosis of A (sum of scores for five parameters: 5-6) will be allowed into this trial
9. Subjects with HBV infection must be on antiviral therapy per regional standard of care guidelines prior to initiation of study therapy. Both HBeAg positive and negative subjects will be included.
10. Patients must have lesions in the liver that are amenable to CT-guided liver biopsy
11. Patients must have normal organ and marrow function as defined below:

    * Haemoglobin ≥ 8.5g/dL
    * Absolute Neutrophil Count ≥ 1.5 x 10^9/L
    * Platelets ≥ 50 x 10^9/L
    * Total Bilirubin < 3 mg/dL
    * AST(SGOT)/ALT (SGPT) ≤ 3 x ULN
    * Creatinine ≤ 1.5 x ULN or measured/calculated Creatinine Clearance (CrCl) ≥ 60 ml/min
12. Ability to understand and the willingness to sign a written informed consent document.
13. Any surgery must be more than 28 days before start of study drug and any surgical wounds must be completely healed
14. Female subjects of childbearing potential must have a negative serum or urine pregnancy test within 3 days prior to receiving the first dose of study medication, and must agree to adequate contraception use from time of signing the informed consent through to 120 days after the last dose of the study drug. Male subjects must agree to adequate contraception use from time of signing the informed consent through 120 days after the last dose of the study drug.

Exclusion Criteria:

1. Patients are excluded if they are receiving any other investigational agents or using an investigational device within 4 weeks of first dose of treatment. Patients are excluded if they are receiving other systemic therapy within 2 weeks of first dose of treatment.
2. Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
3. Prior use of anti-PD1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any drug specifically targeted T-cell costimulatory checkpoint pathways
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension or psychiatric illness/social situations that would limit compliance with study requirements.
5. Subjects with any active autoimmune disease or history of known or suspected autoimmune disease requiring systemic therapy within the past 2 years, except for subjects with vitiligo, resolved childhood asthma/atopy or euthyroid patients with a history of Grave's disease (subjects with suspected autoimmune thyroid disorders must be negative for thyroglobulin and thyroid peroxidase antibodies and thyroid stimulating immunoglobulin prior to randomization). Replacement therapy (e.g. with thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency etc) is not considered a form of systemic treatment
6. Pregnant women or breastfeeding mothers are excluded from this study because of the potential risks to the foetus or baby. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
7. Diagnosis of immunodeficiency, including HIV/AIDS
8. Prior organ allograft or allogeneic bone marrow transplantation
9. History of severe hypersensitivity reactions to other monoclonal antibodies.
10. Prisoners or subjects who are involuntarily incarcerated
11. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness
12. Inability to comply with restrictions and prohibited activities/treatments in this study
13. Chronic treatment with systemic steroids or other immunosuppressive agent.
14. Subjects with concomitant second malignancies (except adequately treated non-melanomatous skin cancers, in situ cervical cancers, localized prostate cancer or in situ breast cancer) are excluded unless a complete remission was achieved at least 3 years prior to study entry and no additional therapy is required or anticipated to be required
15. Prior radiation therapy to the liver or upper abdomen
16. Inability to undergo Y-90 radioembolisation due to inability to cathterise the hepatic artery, portal vein thrombosis/occlusion limiting the ability to perform selective infusion, Tc-99M MAA scan showing unfavourable shunt fraction between the liver and pulmonary parenchyma, any other contraindications to RE as determined by the interventional radiologist (e.g. other anatomic variants precluding safe administration of Y90, severe peripheral vascular disease, uncorrectable coagulopathy etc)

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-12-20 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Response Rate | Tumour assessment at 8 weeks

SECONDARY OUTCOMES:
Time to Response | From date of first dose with Y90 Radioemolization (RE) until best overall response of Complete Response (CR) or Partial Response (PR) is achieved, up to 12 weeks after last dose of Nivolumab
Duration of Response | From date of first assessment of CR or PR until the first date that progressive disease or death is documented, up to 2 years
Time to Progression | From date of first dose with Y90 RE until the first date that progressive disease is documented, up to 12 weeks after last dose of Nivolumab
Progression Free Survival | From date of first dose with Y90 RE until tumour progression, or death from any cause, up to 12 weeks after last dose of Nivolumab
Overall Survival | From date of first dose with Y90 RE until death from any cause, up to 2 years
Quality of Life using the FACT-HEP score | From date of screening until 3 months after last dose of Nivolumab
Quality of Life using EORTC QLQ-C30 | From date of screening until 3 months after last dose of Nivolumab
Adverse events from the combination of RE and nivolumab assessed by NCI CTCAE v4.0 | While receiving study agent and up to 100 days after last dose of Nivolumab

CONTACTS AND LOCATIONS:
Overall Officials: David Wai-Meng TAI, MD, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre - Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tai D, Loke K, Gogna A, Kaya NA, Tan SH, Hennedige T, Ng D, Irani F, Lee J, Lim JQ, Too CW, Ng MCH, Tham CK, Lam J, Koo SL, Chong HS, Goh GB, Huang HL, Venkatanarasimha N, Lo R, Chow PKH, Goh BKP, Chung A, Toh HC, Thng CH, Lim TKH, Yeong J, Zhai W, Chan CY, Choo SP. Radioembolisation with Y90-resin microspheres followed by nivolumab for advanced hepatocellular carcinoma (CA 209-678): a single arm, single centre, phase 2 trial. Lancet Gastroenterol Hepatol. 2021 Dec;6(12):1025-1035. doi: 10.1016/S2468-1253(21)00305-8. Epub 2021 Oct 23. PMID 34695377